CLINICAL TRIAL: NCT04175561
Title: A Dose of Nature: An Interdisciplinary Study of Green Prescriptions and the Environment-Microbiome-Health Axis
Brief Title: A Dose of Nature: An Interdisciplinary Study of Green Prescriptions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sheffield (Other)
Collaborators: Greener Practice, Sheffield (Unknown); Sheffield Network North Primary Care Network (PCN) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRAS 263091
Record Dates: First submitted 2019-11-18; First posted 2019-11-25 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Mental Health Issue; Depression
Keywords: Green prescription; Nature-based health intervention; Nature on prescription; Mental health; Nature connectedness; Nature relatedness; Therapeutic horticulture
MeSH Terms: conditions — Depression; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Social prescribing intervention based on RCT design
Who Masked: Outcomes Assessor
Masking Description: Analytical blinding is possible, but intervention blinding is not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants in the intervention arm will be given a green prescription (gardening activities).
  Interventions: Other: Green prescription
- Control (No Intervention): Participants in the control arm will not be given the intervention.

INTERVENTIONS:
Other: Green prescription — Green prescription intervention will include horticultural activities such as planting, harvesting, learning about ecology and sustainable food growing.
  Arms: Intervention

SUMMARY:
The idea that spending time in natural environments can enhance one's health has been researched for several years. However, the concept of green prescribing--or prescribing a systematic nature-based intervention that can be monitored over time--has only recently generated traction in practice (although the principles can be traced back to several hundred years ago).

Green prescriptions (social prescribing with nature) could potentially help to reduce the costs of mainstream healthcare and could have important 'co-benefits', for example, by simultaneously enhancing the environment.

There are still a number of critical questions that need answering, such as what works best for whom, where and when, and a number of key constraints need to be addressed. The conceptual framework for this proposed trial has been informed by the results of a UK-wide green prescribing questionnaire (Stage 1 of PhD) and recommendations from the Improving Wellbeing through Urban Nature (IWUN) research project (www.iwun.uk).

The main (perceived) constraints to green prescribing acquired from the questionnaire include:

- A lack of funding for all stakeholders

* The research project aims to be cost-effective and not strictly reliant on other organisations

  - A lack of knowledge of how to start a green prescribing service
* The project aims to demonstrate how to start a green prescribing service

  - A lack of opportunities and awareness of service availability
* As above

  - Patient motivation and ease of access/travel etc.
* The novel situational aspect of the project (within the premises of GP practices) aims to maximise access/minimise travel for patients

  - A lack of knowledge of the evidence and mechanisms
* The research project aims to collect evidence on mental health, wellbeing and nature connectedness via an RCT-style experimental design

  - Referral and set-up time
* As per funding objective - see top. The research project will also evaluate patient appointments/attendances (number and frequency) via the RCT approach

The researcher is proposing to conduct a 3-6 month randomised controlled trial (RCT) interventional study involving adult patients with mild-moderate depression as determined using the well-established PHQ-9 questionnaire. A key aim is to sustain this green prescribing service once the research is complete and to hopefully stimulate other trials across Sheffield and the UK (providing opportunities for important meta-analyses).

The intervention will include pocket gardening (activities in small, semi-permanent, versatile gardens) and nature-based activities hosted in the premises of GP surgeries in Sheffield's Network North region.

DETAILED DESCRIPTION:
A green prescription is a prescribed nature-based health intervention designed for individuals with a defined need (or to complement orthodox medical treatments). Common examples of green prescribing activities include: therapeutic horticulture, biodiversity conservation volunteering, care farming, wild crafts and nature walks. Green prescriptions are typically provided for a set length of time (e.g. 12 weeks) but can be open ended.

As a green prescribing activity, therapeutic horticulture has several potential benefits including physical and mental health improvements, facilitating social co-mingling, educational and reward-based e.g. harvesting natural produce. It has already proven successful as a green prescribing activity in projects such as SAGE Greenfingers (sagesheffield.org.uk), which was established following a community needs assessment commissioned by Pitsmoor surgery in Sheffield.

This kind of green prescription provides natural environmental features, social context and meaningful activities - three important interacting phenomena in nature-based interventions. By integrating other nature-based activities such as simply noticing the local wildlife, this project also aims to open pathways (via senses, compassion, emotion meaning and beauty) to nature connectedness - one's emotional relationship with the natural world. The novel situational element of this project (i.e. hosted in GP surgery premises) aims to maximise accessibility and minimise travel for the patients, and to minimise multi-stakeholder logistics.

Furthermore, several policy statements--informed by empirical evidence--were recently published by the IWUN research project (www.iwun.uk). Amongst many other recommendations, these call for GP practices to enhance the biodiversity in their premises.

Importantly, the question of how GP practices can provide their own greenspaces to improve the mental health of their patients is also raised.

Re-designing the outdoor spaces surrounding GP practices and/or integrating new nature-based features and activities within these spaces could help to enhance patient (and staff) wellbeing. Creating pocket gardens (small multifunctional gardens typically installed in the pockets of empty urban spaces) and biodiverse spaces for green prescribing activities is one potential route, and an evaluation of this concept forms the basis of the research project.

There is also a severe lack of randomised controlled trial experiments in green prescribing research - further strengthening the rationale for the chosen experimental approach.

ELIGIBILITY:
Inclusion Criteria:

* Only adults - over 18 years of age with mild-moderate depression.
* Patients will be residents of North Sheffield and part of the Network North Primary Care Network (PCN).
* Patients will preferably be comfortable with outdoors and social settings.

Exclusion Criteria:

* Those who are not adults - over 18 years of age with mild-moderate depression.
* Patients who are not residents of North Sheffield and part of the Network North Primary Care Network (PCN).
* Patients who are not comfortable with outdoors and social settings.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) scale questionnaire assessing change in symptoms of depression | Baseline (start of study), during (at 6 weeks), and post intervention (at 3 months)
  Results of Patient Health Questionnaire-9 scale questionnaire (determining level of depression) will be the primary outcome measure. The PHQ-9 severity cut-off for this study will be as follows:
  * Mild = 5-9
  * Moderate = 10-14 (where a lower score indicates lower level of depression to a minimum score of 5 and a maximum score of 14 for higher levels of depression)

SECONDARY OUTCOMES:
Nature Connectedness Index questionnaire assessing change in level of nature connectedness | Baseline (start of study), during (at 6 weeks), and post intervention (at 3 months)
  Results from the Nature Connectedness Index questionnaire to determine level of nature connectedness. This instrument comprises 6 questions and a 7-point response scale from "completely agree" to "completely disagree" (where 0 is lowest score of nature connectedness and 42 is the maximum score).
Perceived Stress Scale (PSS) questionnaire assessing change in symptoms of stress | Baseline (start of study), during (at 6 weeks), and post intervention (at 3 months)
  Results from the Perceived Stress Scale questionnaire. This is a 10-point measure using a 0-4 Likert style response system.
  Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress. Scores ranging from 0-13 would be considered low stress.
Warwick and Edinburgh Mental Wellbeing Scale (WEMWBS) assessing change in levels of wellbeing | Baseline (start of study), during (at 6 weeks), and post intervention (at 3 months)
  Results from the Warwick and Edinburgh Mental Wellbeing Scale. The Warwick and Edinburgh Mental Wellbeing Scale has 14 x statements and 5 x response categories, summed to provide a single score (where 14 is the lowest score of wellbeing and 70 is the maximum).